CLINICAL TRIAL: NCT07213388
Title: Effects of Different Physical Activity Modalities on Physiological and Psychological Outcomes
Brief Title: Immersive Virtual Reality vs Treadmill Exercise Project
Acronym: IVRTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan University (Other)
Responsible Party: Principal Investigator, Bethany Raiff, Professor, Rowan University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PRO-2023-123
Record Dates: First submitted 2025-02-19; First posted 2025-10-08 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Control; Virtual Reality Physical Activity; Treadmill
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Three group, randomized trial
Masking Description: Participants are not told their group assignment until after completing the pre-session assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Participants will sit quietly while listening to the same music playlist that is played during the VRPA condition.
  Interventions: Behavioral: Control
- Treadmill (Experimental): Participants will walk on a treadmill while listening to the same playlist that is played during the VRPA condition.
  Interventions: Behavioral: Treadmill
- Virtual Reality Physical Activity (VRPA) (Experimental): Participants will wear the VR headset and complete one pre-selected exercise session.
  Interventions: Behavioral: VRPA

INTERVENTIONS:
Behavioral: VRPA — Effects of virtual reality physical activity on outcomes
  Arms: Virtual Reality Physical Activity (VRPA)
Behavioral: Treadmill — Effects of treadmill walking with music on outcomes
  Arms: Treadmill
Behavioral: Control — Effects of music while sitting on outcomes
  Arms: Control

SUMMARY:
The purpose of this research project is to examine the feasibility and acceptability of a virtual reality-based physical activity (VRPA) intervention for inactive adults compared to more traditional forms of physical activity. The project will explore the relationship between VRPA engagement and cognition, biological measures (calories burned, heart rate, and active minutes), rate of perceived exertion, flow, affect, and enjoyment in physical activity as well.

DETAILED DESCRIPTION:
The feasibility and acceptability of a Virtual Reality Physical Activity (VRPA) intervention will be examined. VRPA will be compared with more traditional modes of physical activity (e.g., walking on a treadmill) with regard to physical biomarkers (i.e., heart rate, calories burned, active minutes), flow state (i.e., Flow Short Scale), cognition (e.g., Stroop Test, Trail Making Test, Digital version of the WRAML-2 Symbolic Working Memory Test-Part 1, and Digital Backward Digit Span), affect (e.g., Activation-Deactivation Adjective List and DASS-21), perceived exertion (e.g., Borg's Rate of Perceived Exertion and one question regarding how hard they think they will exert themselves), willingness (i.e., to pay, intent to engage in physical activity), and physical enjoyment (i.e., Physical Activity Enjoyment Scale).

1. Recruit and enroll 60 participants

   a. Participants will be recruited through the SONA system (i.e., student pool for collecting psychological research), word-of-mouth, email lists, flyers, and online classified ads
2. Participants will be screened to ensure they meet the inclusion criteria
3. Participants will be randomly assigned to one of three conditions (VR, Treadmill + Music, Sitting + Music)
4. Participants will complete baseline measures a. Demographic information will be collected (e.g., ethnicity, height, weight, experience with exergames, current physical activity, physical activity readiness) b. Participants will: i. Complete the following surveys

1. Cognition 2. Affect 3. How hard do they think they will exert themselves 4. Willingness ii. Get the following measurements taken:

1. Heart Rate (HR) 6. Participants will engage in a warm-up/acclimation period on either the VR exergame or treadmill condition 7. Participants will engage in exercise for 20-30 minutes in the VR/treadmill condition, or sit quietly listening to music (control condition)

1. HR will be measured during all 3 conditions
2. The treadmill condition will be configured to a level that allows participants to engage in comfortable conversation while experiencing some breathlessness (i.e., brisk/moderate pace) 8. Post-exercise/sitting, participants will

a. Complete the following surveys: i. Feasibility ii. Acceptability iii. Cognition iv. Flow v. Affect vi. Borg's Rate of Perceived Exertion (RPE) vii. Willingness viii. Physical Enjoyment b. Get the following measurements taken: i. Heart Rate ii. Calories burned

ELIGIBILITY:
Inclusion Criteria:

1. Be inactive (i.e., do not meet physical activity guidelines)
2. have no current neurological, psychiatric, sensory, or motor impairment, and normal or corrected-to-normal vision (only thin wire glasses or contacts can be used)
3. have no history of motion sickness
4. have the ability to exercise based on the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) (Warburton et al., 2019)
5. Have not fallen to the point of injury in the last 6 months.
6. Be willing to wear an activity tracker
7. 18-64 years,

Exclusion Criteria:

1. Do not meet the inclusion criteria
2. Struggle to use operate a VR headset
3. Cannot read
4. Have concerns about balance/falling while using a VR headset,
5. Unable to provide informed consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Pace of participant recruitment | Up to 24 months
  enrollment rate of 6 participants per month
Number of participants willing to continue using the assigned exercie modality | Day 1
  Willingness to continue using the exercise modality to which the participants were assigned and self-report enjoyment from engaging in the assigned exercise.
Percentage of participants who complete the required tasks in each condition | Day 1
  Are participants able to complete the required tasks

SECONDARY OUTCOMES:
Changes in Heart Rate | Day 1
  Differences in heart rate from pre- to post session
Self-reported measures of "flow" associated with the assigned conditions | Day 1
  Flow will be assessed using the Flow Short Scale (Rheinberg et al, 2003) that is comprised of 13 questions answered on a 7-point scale (1 = Not at all, 7 = very much). Scores can range from 13-91, with lower scores indicating less of a "flow state" or feelings of immersion in the assigned activity.
Changes in affect | Day 1
  Using the Activation-Deactivation Checklist (Thayer et al., 1986), participants will rate 20 different adjectives on a 4-point scale (1= definitely feel, 2= feel slightly, 3= cannot decide, 4= definitely do not feel) before they engage in the assigned activity and after they engage in the assigned activity. Lower numbers will indicate higher endorsements of a particular feeling, but the primary outcome will examine any changes in pre- to post-activity ratings of the different affective states.
Rate of percieved exertion | Day 1
  Borg's Rate of Perceived Exertion will be used to measure how participants rate their perceived exertion on a scale of 6 (no exertion at all) to 20 (maximal exertion) (Borg, 1982). The scale is anchored to the participant's subjective perception, with descriptors such as "extremely hard." Rate of perceived exertion will be evaluated post-activity only and will be compared across groups.
Changes in Stroop Color and Word Test | Day 1
  The Stroop Color and Word Test (Golden et al, 2002) will be conducted pre- and post-assigned activities. Raw scores (e.g., reaction times, errors) will be calculated and changes in those scores from pre- to post-activity will be determined.
Number of Calories Burned | Day 1
  Total number of calories burned during the assigned condition
Number of Active Minutes | Day 1
  Total number of active minutes during the assigned condition
Changes in Executive Functioning | Day 1
  The Trail Making Test (TMT) will be used to calculate changes in executive function (Arbuthnott & Frank, 2000; Kortte et al., 2002; Reitan, 1956). Participants will be required to draw lines connecting different scattered numbers (Part A) and scattered numbers and letters (Part B). If the test can not be completed in 5-minutes it will be stopped. The more errors a person makes, and the longer a person takes, indicate poorer outcomes for executive function and changes in this measure will be calculated from pre- to post-activity.
Changes in Working Memory Capacity | Day 1
  The Backward Digits Span (BDT, Lamar et al., 2007) measures an individual's working memory capacity and is comprised of 21 trials where participants will need to recall 3, 4, and 5-digit spans. The more numbers a person can correctly recall the better their working memory. Changes in this measure, from pre- to post-activity, will be calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Rowan University, Glassboro, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers can request deidentified data sets after the research team has published all planned analyses related to this research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: September 2026 until August 2036
Access Criteria: Researchers will be able to access the data upon request. The PI will securely share the requested IPD.